CLINICAL TRIAL: NCT06463093
Title: Contribution of Brain Positon Emission Tomography With 18 Flurodeoxyglucose Labelled With Fluorine 18 for the Differential Diagnosis of Cognitive Disorders of Psychiatric or Neurodegenerative Origin
Brief Title: Differential Diagnosis of Cognitive Disorders of Psychiatric or Neurodegenerative Origin
Acronym: ATEPDIPSY
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Antoine VERGER, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2023PI120
Record Dates: First submitted 2023-11-27; First posted 2024-06-17 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Neurocognitive Disorders
MeSH Terms: conditions — Neurocognitive Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the research is to analyze whether 18F-FDG PET helps in the diagnosis and therefore in the management of the patient.

DETAILED DESCRIPTION:
Neurocognitive disorder or Mild Cognitive Impairment corresponds to a decline in one or more cognitive functions; compared to the previous level of performance.

Indeed, the prevalence of neurodegenerative pathologies is estimated at more than one million according to Santé Publique France, due to the aging of the population. To be compared with the prevalence of the population suffering from a psychiatric disorder estimated at one in five people, or 13 million French people, in 2021.

With the increase in the prevalence of these two entities and their clinical entanglement, the question arises of the origin of neurocognitive disorders, is it a manifestation of a psychiatric pathology or a neurodegenerative pathology not yet diagnosed.

If this is the case, the patient's prognosis is modified with a pejorative evolution and a loss of autonomy which is to be anticipated. This delay deprives the patient and his family of interventions likely to alleviate behavioral disorders; maintain a level of autonomy compatible with life at home; alleviates the burden and improves the quality of life of caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with cognitive impairment
* Positron emission tomography with flurodeoxyglucose labeled with fluorine 18 carried out in the course of care

Exclusion Criteria:

* Patients objecting to the collection of their data

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for psychiatric reasons with neurocognitive disorders in the clinic, having consulted or being hospitalized at the psychotherapeutic center of Nancy between 01/01/2021 to 01/01/2024 and having undergone a flurodeoxyglucose positron emission tomography marked with fluorine 18 carried out in the course of care
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-11-30 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-07-02 (Estimated)

PRIMARY OUTCOMES:
Neuro cognitive disorders and disorders of neurodegenerative origin in psychiatric population | one day
  Change of the diagnosis before the PET and after the PET

CONTACTS AND LOCATIONS:
Locations (1):
- Nancy's hospital, Vandœuvre-lès-Nancy, France